CLINICAL TRIAL: NCT06897241
Title: Personalized Metabolic Responses to Rapid, Slow and Resistant Starch (PerStarch)
Brief Title: Personalized Metabolic Responses to Rapid, Slow and Resistant Starch
Acronym: PerStarch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Federico II University of Naples, Department of Clinical Medicine and Surgery, Naples, Italy (Unknown); Göteborg University (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PerStarch
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Adults With Overweight and Obesity
Keywords: Glucose metabolism; Prevotella; AMY1 copy number; Continuous glucose monitoring; Meal tolerance test; Fecal redox potential; Home sampling
MeSH Terms: conditions — Obesity | interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: Three-way cross-over design, where subjects are randomized to the order of the three different interventions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Resistant starch (Experimental): Participants will consume 80 grams of carbohydrates from resistant starch during the meal challenges and two times daily during the 14-day intervention period
  Interventions: Other: Resistant starch; Other: Slow digestible starch; Other: Rapid digestible starch
- Slow digestible starch (Active Comparator): Participants will consume 80 grams of carbohydrates from slow digestible starch during the meal challenges and two times daily during the 14-day intervention period
  Interventions: Other: Resistant starch; Other: Slow digestible starch; Other: Rapid digestible starch
- Rapid digestible starch (Other): Participants will consume 80 grams of carbohydrates from rapid digestible starch during the meal challenges and two times daily during the 14-day intervention period
  Interventions: Other: Resistant starch; Other: Slow digestible starch; Other: Rapid digestible starch

INTERVENTIONS:
Other: Resistant starch — Participants will consume 80 grams of carbohydrates from resistant starch during the meal challenges and two times daily during the 14-day intervention period
Other: Slow digestible starch — Participants will consume 80 grams of carbohydrates from slow digestible starch during the meal challenges and two times daily during the 14-day intervention period
Other: Rapid digestible starch — Participants will consume 80 grams of carbohydrates from rapid digestible starch during the meal challenges and two times daily during the 14-day intervention period

SUMMARY:
The study aims to investigate how individuals with varying gut microbiota composition and AMY1 gene copy number respond to three different types of starch. A 12-week trial will therefore be conducted, where all participants will go through three different 17-day interventions in a randomized order. Each intervention will contain a different type of starch:

A) Resistant starch B) Slow digestible starch C) Rapid digestible starch

Each intervention will contain a preparation day, a meal challenge test day at clinic, a 14-day dietary intervention at home followed by a follow up visit at clinic. The interventions will be separated with a 14-day wash-out period, where participants are consuming their normal food.

Blood, saliva and fecal samples will be collected during the trial, together with data from continuous glucose monitoring and body measurements. Questionnaires on dietary intake and lifestyle, food preferences, self-reported appetite, health-related quality of life, sleep quality and daytime sleepiness will also be filled out by the participants.

DETAILED DESCRIPTION:
Up to 400 men and women with overweight or obesity will be invited for screening. Participants will provide stool-, saliva-, and fasting blood samples, alongside undergoing anthropometric measurements. Gut microbiota will be analyzed from stool samples, while saliva samples will be used to determine AMY1 copy number. This data will then be used to categorize participants into four distinct groups, based on high or low Prevotella abundance and high or low AMY1 copy number.

Participants in all four groups will undergo a three-way cross-over feeding regime containing three different types of starch: A) resistant starch (RS), B) slow digestible starch (SDS) and C) rapid digestible starch (RDS). Each treatment will start with a "meal challenge day" at the clinic, where participants will eat test foods for breakfast, containing the different types of starch, followed by a standardized lunch. During the meal challenge day, blood samples will be collected over 7 hours along with continuous glucose monitoring, saliva sampling and self-reported appetite. During the following 14 days, participants will continue to consume the test foods A, B or C for lunch and dinner at home along with continuous glucose monitoring. The at home intervention will be followed up with a clinical visit, where fasting blood samples are taken before the breakfast from the meal challenge day is repeated. After the breakfast, participants will take finger prick blood samples from home during another 4 hours. Each intervention will be followed by a 14-day wash out period before the next treatment begins.

The specific aims with the trial are:

1. To investigate differential metabolic responses (glycemia, blood lipids and inflammation biomarkers) in response to meal tolerance tests based on RS, SDS or RDS served for breakfast and dinner across individuals with high or low abundance of Prevotella and high or low AMY1 copy number.
2. To evaluate metabolic effects of chronic consumption of RS and SDS versus RDS daily for two weeks across different enterotypes and in individuals with high or low AMY1 copy number.
3. To evaluate a non-invasive method to measure redox potential in fecal samples. In exploratory analyses, the associations between fecal redox potential and responses to different starches as well as microbiota and other biomarkers will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopausal women
* Age 30-75 years
* BMI 27-40 kg/m2
* Waist circumference > 102/88 cm for men/women
* Weight stable during previous 3 months (± 3 kg)
* Willingness to consume the intervention diets
* Ability to deal with the monitoring devices
* Medications stable for the previous 14 days
* Signed informed consent

Exclusion Criteria:

* Cardiovascular events (myocardial infarction or stroke) during the previous 6 months
* Diagnosis of diabetes (any type) or use of any drug who can interfere with glucose homeostasis (i.e., metformin, incretin analogues, SGLT-2 inhibitors)
* History of stomach or gastrointestinal conditions (inflammatory bowel disease, Crohn's disease, malabsorption, etc.)
* Colostomy, bowel resection, bariatric surgery or other major gastrointestinal surgery
* Renal or liver failure (creatinine <1.7 mg/dl and alanine aminotransferase/aspartate aminotransferase < 2 times than normal values, respectively)
* Anemia (hemoglobin below the age and sex specific normal reference ranges at screening)
* Blood donation (or participation in a clinical study with blood sampling) within 30 days prior to inclusion
* Having been treated with antibiotics within the past 3 months or planning to undergo treatment during the study period.
* Habitual use of probiotic/prebiotic supplements or foods enriched in probiotics
* Celiac disease
* Vegan/vegetarian diet (or a diet incompatible with protocol diets)
* Intense physical activity regimen (> 7 h/week of moderate intensity or > 3 h/week of high intensity)
* History of drug or alcohol abuse
* Not able to understand written and spoken Swedish
* Any other reason for lack of suitability for participation in the trial, as judged by the principal investor or co-principal investigator

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Propionate | During meal challenge day (at the beginning of each intervention)
  Differences in plasma propionate between strata at timepoint +360 min

SECONDARY OUTCOMES:
Glucose (7 h, between treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in glucose responses (from 7-hour meal challenge test) between dietary treatments during whole day for all participants
Insulin (7 h, between treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in insulin responses (from 7-hour meal challenge test) between dietary treatments during whole day for all participants
Glucose (7 h, within treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in glucose responses (from 7-hour meal challenge test) across strata within the same dietary treatment
Insulin (7 h, within treatments) | During meal challenge day (at the beginning of each intervention)
  Differences insulin responses (from 7-hour meal challenge test) across strata within the same dietary treatment
Glucose (4 h, breakfast, between treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in glucose between dietary treatments during breakfast meals separately for all participants
Insulin (4 h, breakfast, between treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in insulin between dietary treatments during breakfast meals separately for all participants
Glucose (4 h, breakfast, within treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in glucose during breakfast meals separately across strata within the same dietary treatment
Insulin (4 h, breakfast, within treatments) | During meal challenge day (at the beginning of each intervention)
  Differences in insulin responses during breakfast meals separately across strata within the same dietary treatment
CGM (between treatments) | During each intervention (14 days)
  Differences in 24-hour CGM-measures and in the dynamic features of the postprandial glucose response as evaluated by CGM-home sampling between dietary treatments for all participants
CGM (within treatments) | During each intervention (14 days)
  Differences in 24-hour CGM-measures and in the dynamic features of the postprandial glucose response as evaluated by CGM-home sampling between strata within dietary treatment
Glucose (home sampling) | Att the end of each 14-day intervention
  Differences in glucose from home sampling between dietary treatments for all participants
C-peptide (home sampling) | At the end of each 14-day intervention
  Differences in C-petide from home sampling between dietary treatments for all participants
CRP | During meal challenge test (at the beginning of each intervention)
  Differences in inflammation biomarkers (CRP) between dietary treatments for all participants
Blood lipids | During each intervention (meal challenge test and home sampling)
  Differences in blood lipids between dietary treatments for all participants
Short chain fatty acids | During each intervention (fasting samples and meal challenge test)
  Differences in short chain fatty acids (from feces and plasma) between dietary treatments for all participants

OTHER OUTCOMES:
Metabolomics | During meal challenge day (at the beginning of each intervention)
  Differences in metabolomics from 7-hour meal challenge test between dietary treatments for all participants
GLP-1 | During meal challenge day (at the beginning of each intervention)
  Differences in GLP1 from 7-hour meal challenge test between dietary treatments for all participants
GIP | During meal challenge day (at the beginning of each intervention)
  Differences in GIP from 7-hour meal challenge test between dietary treatments for all participants
Anthropometry | During each intervention (14 days)
  Differences in anthropometric measures between dietary treatments for all participants
Sleep quality | During each intervention (14 days)
  Differences in sleep quality between dietary treatments for all participants (measured with Pittsburgh Sleep Quality Index). The result is presented as a global sleep score on a 0-21 scale. A higher score indicates worse sleep quality and a value > 5 is classified as "poor sleep". For the areas subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction, component scores can also be calculated, each on a 0-3 AU scale.
Daytime sleepiness | During each intervention (14 days)
  Differences in daytime sleepiness between dietary treatments for all participants (measured with Epworth Sleepiness Scale). The result is presented as an ESS-score on a 0-24 scale, where a higher score indicates greater daytime sleepiness. A value > 10 is classified as excessive daytime sleepiness.
Health-related quality of life | During each intervention (14 days)
  Differences in health-related quality of life between dietary treatments for all participants (measured with SF-36v2). Domain scores are calculated for the areas physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional health and mental health. These can be presented either on a 0-100 scale of arbitrary units (raw scores) or as a norm-based T-score (with a mean of 50 AU and a standard deviation of 10). A higher score indicates greater HRQoL. T-scores are also calculated for the aggregated dimensions of physical- and mental health.
Self-reported appetite | During meal challenge test (at the beginning of each intervention)
  Differences in self-reported appetite between dietary treatments for all participants (measured with visual analogue scales). Participants will assess subjective feelings of appetite such as hunger, desire to eat and fullness by marking on a 100 mm scale with end descriptions ranging from "Not at all" (0) to "Extremely" (100).
Fecal redox potential and metabolic responses | During each intervention (14 days)
  Associations between fecal redox potential and responses to different starches
Fecal redox potential and microbiota | During each intervention (14 days)
  Associations between fecal redox potential and microbiota
Fecal redox potential and clinical biomarkers | At baseline
  Associations between fecal redox potential and clinical biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Principal Investigator — Chalmers University of Technology
Locations (1):
- Clinical Trial Center, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided